CLINICAL TRIAL: NCT00630292
Title: Feasibility Study of Vessel Analysis for Noninvasive Diagnosis of Malignancy in Breast Tumors
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Existing vessel analysis software could not be applied to breast MRI data.
Sponsor: University of North Carolina, Chapel Hill (Other)
Responsible Party: Lisa Carey/ Principal Investigator, University of North Carolina-Chapel Hill
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: LCCC0718
Record Dates: First submitted 2008-02-28; First posted 2008-03-07 (Estimated); Results first posted 2010-05-05 (Estimated); Last update posted 2010-05-18 (Estimated); Status verified 2010-05

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — tocilizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Other: Magnetic Resonance Angiography (MRA) of the Breast

INTERVENTIONS:
Other: Magnetic Resonance Angiography (MRA) of the Breast — Magnetic Resonance Angiography (MRA) of the breast will be performed before or after pre-treatment magnetic resonance imaging (MRI) and then once again before or after the post-treatment MRI.

SUMMARY:
This is a pilot study designed to explore the feasibility of non-invasively diagnosing the presence of cancer in the breast using non-invasive magnetic resonance imaging (MRI) methods and an analysis of vessel shape defined from these magnetic resonance images.

ELIGIBILITY:
Inclusion Criteria:

* adult women (age >= 18),
* with Histologically documented newly diagnosed stage II-IV invasive breast cancer appropriate for neoadjuvant (preoperative) systemic therapy.
* ECOG performance status of 0, 1, or 2 at the initiation of the study.

Exclusion Criteria:

* pregnant women
* women with contralateral mastectomies
* known bilateral tumors
* subjects prone to claustrophobia
* contraindicated to have MRI
* mentally impaired
* not fluent in english

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2008-03; Primary Completion 2008-12 (Actual); Study Completion 2009-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Irvin, MD, Principal Investigator — UNC-CH
Locations (1):
- UNC Hospitals, Chapel Hill, North Carolina, United States

REFERENCES:
- [Background] Pisano ED, Gatsonis C, Hendrick E, Yaffe M, Baum JK, Acharyya S, Conant EF, Fajardo LL, Bassett L, D'Orsi C, Jong R, Rebner M; Digital Mammographic Imaging Screening Trial (DMIST) Investigators Group. Diagnostic performance of digital versus film mammography for breast-cancer screening. N Engl J Med. 2005 Oct 27;353(17):1773-83. doi: 10.1056/NEJMoa052911. Epub 2005 Sep 16. PMID 16169887
- [Background] Kriege M, Brekelmans CT, Boetes C, Besnard PE, Zonderland HM, Obdeijn IM, Manoliu RA, Kok T, Peterse H, Tilanus-Linthorst MM, Muller SH, Meijer S, Oosterwijk JC, Beex LV, Tollenaar RA, de Koning HJ, Rutgers EJ, Klijn JG; Magnetic Resonance Imaging Screening Study Group. Efficacy of MRI and mammography for breast-cancer screening in women with a familial or genetic predisposition. N Engl J Med. 2004 Jul 29;351(5):427-37. doi: 10.1056/NEJMoa031759. PMID 15282350
- [Background] Thukral A, Thomasson DM, Chow CK, Eulate R, Wedam SB, Gupta SN, Wise BJ, Steinberg SM, Liewehr DJ, Choyke PL, Swain SM. Inflammatory breast cancer: dynamic contrast-enhanced MR in patients receiving bevacizumab--initial experience. Radiology. 2007 Sep;244(3):727-35. doi: 10.1148/radiol.2443060926. PMID 17709827
- [Background] McDonald DM, Baluk P. Significance of blood vessel leakiness in cancer. Cancer Res. 2002 Sep 15;62(18):5381-5. PMID 12235011
- [Background] Bullitt E, Reardon DA, Smith JK. A review of micro- and macrovascular analyses in the assessment of tumor-associated vasculature as visualized by MR. Neuroimage. 2007;37 Suppl 1(Suppl 1):S116-9. doi: 10.1016/j.neuroimage.2007.03.067. Epub 2007 Apr 25. PMID 17512217
- [Background] Bullitt E, Zeng D, Gerig G, Aylward S, Joshi S, Smith JK, Lin W, Ewend MG. Vessel tortuosity and brain tumor malignancy: a blinded study. Acad Radiol. 2005 Oct;12(10):1232-40. doi: 10.1016/j.acra.2005.05.027. PMID 16179200
- [Background] Bullitt E, Wolthusen PA, Brubaker L, Lin W, Zeng D, Van Dyke T. Malignancy-associated vessel tortuosity: a computer-assisted, MR angiographic study of choroid plexus carcinoma in genetically engineered mice. AJNR Am J Neuroradiol. 2006 Mar;27(3):612-9. PMID 16552004

RESULTS

PARTICIPANT FLOW:
Groups:
- Breast Magnetic Resonance Angiography: Women who had a Magnetic Resonance Angiography sequence added to a clinical breast MRI
Period: Overall Study
Arm/Group | Breast Magnetic Resonance Angiography
Started | 6
Completed | 5
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Breast Magnetic Resonance Angiography
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 1
Age Continuous [Mean (Standard Deviation); unit: years] | 45.5 (5.49)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Amount of Blood Vessel Tortuosity in Breast With Known Cancer
Description: Amount of vessel tortuosity before the start of neoadjuvant chemotherapy and at the end of neoadjuvant chemotherapy
Time Frame: up to two weeks prior to start of chemotheraphy
Population: Blood vessels could not be detected for any of the subjects due to spatial resolution limits of MRI scanner for breast MRI and therefore measurement of blood vessel angularity could not be performed.
Measure: Number; unit: sum of blood vessel angles
Arm/Group | Breast Magnetic Resonance Angiography
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Description: No adverse events were observed.
Arm/Group | Breast Magnetic Resonance Angiography
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

LIMITATIONS AND CAVEATS:
The software used to perform breast vessel analysis failed to detect any vessels in the breast due to the limited spatial resolution possible for breast imaging with the 1.5T Magnetic Resonance Imaging System used in the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes